CLINICAL TRIAL: NCT07293442
Title: Effects of Pelvic Floor Muscle Exercise on Lower Urinary Tract Symptoms, Postvoid Residual Volume and Quality of Life in Patients Undergoing Surgery for Benign Prostatic Hyperplasia.
Brief Title: Pelvic Floor Muscle Exercise for Lower Urinary Tract Symptoms After Surgery for Benign Prostatic Hyperplasia.
Acronym: BPH LUTS PFME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chun Lin, Principal Investigator, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N202511003; 113-WF-IR-10 (Other Grant/Funding Number: Wan Fang Hospital Holistic Care Project Grant)
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: LUTS, Quality of Life
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, parallel-group, randomized controlled trial. Participants will complete a baseline (preoperative) assessment before surgery. After the baseline assessment, participants will be randomly assigned to either the intervention group or the control group.
  Outcome assessments will be conducted at postoperative week 1, week 4, and week 8.
  The study evaluates the effects of pelvic floor muscle exercise on lower urinary tract symptoms, postvoid residual volume, and quality of life following surgery for benign prostatic hyperplasia.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor was blinded. Participants and care providers could not be blinded due to the nature of the pelvic floor muscle exercise intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1：Intervention Group (Pelvic Floor Muscle Exercise Group) (Experimental): Participants in this group will receive a structured pelvic floor muscle exercise (PFME) program.The exercise program is administered after the baseline preoperative assessment and continues through postoperative week 1, week 4, and week 8 follow-up assessments.
  Interventions: Behavioral: pelvic floor muscle exercises
- Arm 2：Control Group (Usual Care Group) (No Intervention): Participants in this group will receive standard perioperative care without pelvic floor muscle exercise training. Baseline preoperative assessments and postoperative follow-ups at week 1, week 4, and week 8 will be conducted in the same schedule as the intervention group.

INTERVENTIONS:
Behavioral: pelvic floor muscle exercises — Participants assigned to the experimental arm will begin pelvic floor muscle exercises (PFME) before undergoing prostate surgery. The preoperative training includes instruction on correct pelvic floor muscle contraction techniques. After surgery, PFME is resumed one week post-operation when hematuria has resolved and continues for four weeks.
  Throughout the intervention period, participants receive regular guidance, exercise log monitoring, and support through a designated LINE communication group. PFME aims to improve lower urinary tract symptoms, reduce postvoid residual volume, and enhance quality of life.
  Arms: Arm 1：Intervention Group (Pelvic Floor Muscle Exercise Group)

SUMMARY:
This study aims to evaluate the effectiveness of pelvic floor muscle exercise (PFME) on improving lower urinary tract symptoms (LUTS), postvoid residual volume (PVR), and quality of life in patients undergoing surgery for benign prostatic hyperplasia (BPH). Patients who undergo BPH-related procedures, such as TURP or HoLEP, often experience postoperative symptoms including urinary urgency, frequency, nocturia, dribbling, and voiding difficulty, which may negatively affect daily living. Pelvic floor muscle exercise is believed to enhance urethral sphincter function and pelvic floor support, thereby improving urinary control. This randomized study assigns participants to either an intervention group receiving PFME training or a control group receiving standard postoperative care. Differences in urinary outcomes between groups will be compared. The findings are expected to provide an accessible and cost-effective rehabilitation strategy to support postoperative recovery and quality of life.

DETAILED DESCRIPTION:
Patients undergoing surgery for Benign Prostatic Hyperplasia (BPH) frequently experience postoperative lower urinary tract symptoms (LUTS), voiding difficulties, urinary incontinence, and reduced quality of life. Pelvic Floor Muscle Exercise (PFME) has been shown to improve pelvic floor strength and urinary function; however, evidence regarding its effectiveness when applied as an early postoperative intervention remains limited. This study uses a pretest-posttest randomized design. All participants undergo baseline assessments before surgery, including LUTS questionnaires, postvoid residual measurement, and quality-of-life evaluation. After baseline assessment, participants are randomly assigned to either group using block randomization.

The intervention group receives standard postoperative care plus PFME training, which includes proper pelvic floor muscle contraction techniques, transversus abdominis coordination training, and the Knack maneuver. Training instruction and demonstrations are provided by the research team. The control group receives standard postoperative care and routine education only. Outcome assessments are conducted at 1 week, 4 weeks, and 8 weeks after surgery to evaluate the impact of PFME on LUTS, voiding function, and quality of life. This study aims to provide evidence for an effective early rehabilitation strategy to enhance postoperative urinary recovery and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older.
2. Diagnosed with benign prostatic hyperplasia (BPH) and scheduled to undergo their first prostate surgery.
3. Able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. Patients with prostate cancer, bladder tumors, or other concomitant urological diseases.
2. Patients with long-term indwelling urinary catheters or suprapubic cystostomy.
3. Patients currently participating in other urology-related clinical trials.

Ages: 18 Months to 99 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Baseline, postoperative week 1, week 4, week 8
  Measures change in lower urinary tract symptoms using the International Prostate Symptom Score (IPSS). Participants complete the IPSS questionnaire at baseline (pre-surgery), and at postoperative week 1, week 4, and week 8.

SECONDARY OUTCOMES:
Change in Postvoid Residual Volume (PVR) | Baseline, postoperative week 1, week 4, week 8
  Postvoid residual urine volume is measured using a non-invasive bladder scanner at baseline (pre-surgery), and at postoperative week 1, week 4, and week 8.
Change in Urinary Incontinence Severity (ICIQ-UI Short Form) | Baseline, postoperative week 1, week 4, week 8
  Urinary incontinence severity is assessed using the ICIQ-UI Short Form questionnaire at baseline, postoperative week 1, week 4, and week 8.
Change in Quality of Life (ICIQ-LUTSqol) | Baseline, postoperative week 1, week 4, week 8
  Quality of life is measured using the ICIQ-LUTSqol questionnaire at baseline, postoperative week 1, week 4, and week 8.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University - Wan Fang Hospital, Taipei
  - Wan Fang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No